CLINICAL TRIAL: NCT01229826
Title: Magnetic Resonance Elastography (MRE) of Uterine Fibroids
Acronym: MRE
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, David A. Woodrum, David A. Woodrum, M.D., PhD., Mayo Clinic
Other Study IDs: 10-002112; Mayo Clinic (Other: Internal Funding)
Record Dates: First submitted 2010-10-22; First posted 2010-10-28 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2015-09

CONDITIONS: Uterine Fibroids
Keywords: Uterine fibroids; Uterine leiomyomas; MR Elastography; MRI (Magnetic Resonance Imaging); Symptomatic Uterine Fibroids
MeSH Terms: conditions — Leiomyoma; Myofibroma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Radiation: MR Elastography — MRE is performed at the end of the examination after the standard MRI protocol. A test vibration is first applied on the patient to familiarize the patient with the vibration. The MRE sequence is performed with either a body coil or a pelvic-array coil. The total acquisition time is split into four periods of suspended respiration of 16 seconds for acquisition of wave images at four phase offsets. To obtain a consistent position of the fibroid for each phase offset, patients are asked to quietly breath and remain still.
  Other Names: Signa; GE Healthcare

SUMMARY:
The purpose of this study is to gain additional information regarding use of Magnetic Resonance Elastography (MRE) for uterine fibroid characterization. In this study, the investigators will use a new noninvasive technology, MRE, to further characterize the elastic properties of the uterine fibroids. To date, very little is known concerning how the tissue composition of the uterine fibroid may affect its treatment with Magnetic Resonance Guided Focused Ultrasound (MRgFUS).

In this study, the investigators will use a new noninvasive technology, magnetic resonance elastography (MRE), to further characterize the elastic properties of the uterine fibroids. This information will be gathered during routine magnetic resonance imaging for symptomatic uterine fibroids. It is known that some fibroids with increased T2-signal on Magnetic Resonance Imaging(MRI) can be more difficult to treat.

This information will be gathered during routine magnetic resonance imaging for symptomatic uterine fibroids.

DETAILED DESCRIPTION:
This is a single-site, non-randomized pilot study to determine whether Magnetic Resonance Elastography (MRE) can be optimized for clinical use as part of the patients routine clinical imaging and to correlate with MR signal characteristics of the uterine fibroid.

MRE is performed at the end of the examination after the standard Magnetic Resonance Imaging protocol.

Aims:

Specific Aim 1: To acquire magnetic resonance elastography images on women who have a clinically ordered pelvic magnetic resonance imaging (MRI) for uterine fibroids.

Specific Aim 2: To examine the correlation between MRE stiffness values and MR T2 signal characteristics for uterine fibroids. For a subset of patients going on to surgery correlation with pathology can also be performed.

This study will seek to determine whether MRE can be performed in the pelvis on a routine clinical basis as well as correlating the MRE findings with magnetic resonance signal characteristics. There are no additional risks to the patient and no additional cost to the MRI exam.

ELIGIBILITY:
Inclusion Criteria:

1. Women able to give informed consent
2. Women having uterine imaging

Exclusion Criteria:

1. Women currently pregnant
2. Allergy to either gadolinium or iodinated contrast
3. Severe claustrophobia
4. Weight in excess of 250 pounds

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Female individuals between the years of 18 and 65 whose doctor has suggested magentic resonance imaging of the uterus for treatment of uterine fibroids.
Sampling Method: Non-Probability Sample
Enrollment: 134 (Actual)
Dates: Start 2010-10; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Acquisition of MR elastography images for comparison. | every six months
  MRE is performed at the end of the examination after the standard Magnetic Resonance Imaging(MRI) protocol.

SECONDARY OUTCOMES:
Examination of Magnetic Resonance Elastography stiffness values and MR T2. | every six months
  To examine the correlation between MR elastography stiffness values and MR T2 signal characteristics for uterine fibroids. For a subset of patients going on to surgery correlation with pathology can also be performed.

CONTACTS AND LOCATIONS:
Overall Officials: David A. Woodrum, M.D., PhD., Principal Investigator — Mayo Clinic - Rochester, Minnesota
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States